CLINICAL TRIAL: NCT02017431
Title: Strengthening the Case for Ongoing Reduction of Exposure to Traffic-Related Air Pollution
Brief Title: Air Pollution and Allergens - Attenuation of Health Effects Particle Reduction
Acronym: DE3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Christopher Carlsten, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: H11-01831/2013
Record Dates: First submitted 2013-12-16; First posted 2013-12-20 (Estimated); Last update posted 2017-09-29 (Actual); Status verified 2017-09

CONDITIONS: Allergies
Keywords: Diesel exhaust; Particle depleted diesel exhaust; Air pollution; Airway responsiveness; Allergies
MeSH Terms: conditions — Hypersensitivity | interventions — Allergens; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Filtered air (Active Comparator): Exposure for 2 hours to filtered air followed by subject specific inhaled allergen challenge
  Interventions: Other: Allergen
- Diesel exhaust (Experimental): Exposure for 2 hours to diesel exhaust followed by subject specific inhaled allergen challenge
  Interventions: Other: Allergen
- Filtered air control (Active Comparator): Exposure for 2 hours to filtered air followed by inhaled saline challenge
  Interventions: Other: Saline
- Particle depleted diesel exhaust (Experimental): Exposure for 2 hours to particle depletion diesel exhaust followed by inhaled allergen challenge
  Interventions: Other: Allergen; Other: Particle depleted diesel exhaust

INTERVENTIONS:
Other: Allergen — Subject specific allergen is inhaled on day 1 of the triad
  Arms: Diesel exhaust; Filtered air; Particle depleted diesel exhaust
Other: Saline — Saline is inhaled on day 1 of the triad
  Arms: Filtered air control
Other: Particle depleted diesel exhaust — High-efficiency particulate filtration of diesel exhaust
  Arms: Particle depleted diesel exhaust

SUMMARY:
The study probes the effects of combined exposures to diesel exhaust and allergens on lung function and on the immune system, specifically focusing on the ability of a particle depletion technique to attenuate effects we and others have seen previously. Individuals are exposed to either filtered air (FA), carefully controlled levels of diesel exhaust (DE) or particle-depleted diesel exhaust (PDDE) in our exposure chamber, after which the investigators will administer an inhaled allergen challenge. 48h later, a procedure called bronchoscopy is used to collect samples from the lungs. After 1 month, the entire procedure is to be repeated with one of the alternate exposures. This will be repeated 4 times (4 exposures; 2 filtered air, 1 diesel exhaust, 1 particle-depleted diesel exhaust)

DETAILED DESCRIPTION:
1. Purpose/Objective:

   The aim of this study is to investigate the ability of depletion of diesel exhaust particles to attenuate adverse effects of diesel exhaust on lung function and on allergic responses.
2. Hypotheses:

   Hypothesis 1: Allergen-specific immune response (specific IgG4, etc; relevant responses in DNA methylation and proteomics) in allergen-challenged airways in sensitized individuals is increased by diesel exhaust "synergy".

   Hypothesis 2: Synergistic responses will be greater in asthmatics than in non-asthmatics.

   Hypotheses 3: Synergy is attributable to the particulate fraction of DE (i.e. is normalized by particle depletion).
3. Justification:

   Diesel exhaust consists of both gaseous and particulate air pollutants. In recent studies, cardiovascular effects seem attenuated when the particulate portion is removed. We would like to know if that is true for respiratory and immunological endpoints. Understanding these changes may help us prevent health problems associated with air pollution in the future.
4. Research Method:

Blinded crossover experiment between four conditions (DE and allergen, PDDE and allergen, FA and allergen, FA and saline), randomized and counter-balanced to order. Each condition will be separated by a 4-week washout period.

An inhaled allergen or saline challenge is delivered after each exposure (DE, PDDE, or FA). 24 h post challenge, airway reactivity will be assessed with a methacholine challenge. 48 h post challenge, bronchoalveolar lavage (BAL), airway brushes and tissue biopsies will be obtained for analysis of immune activation. Nasal lavage samples will also be collected to examine responses in the upper airways and blood and urine will be studied to examine systemic responses. Spirometry and methacholine challenge will be used to assess effects on airway function.

ELIGIBILITY:
Inclusion Criteria:

* Age between 19 and 49 years
* Non-smoking
* Positive skin prick test for at least one of: birch, grass, or dust

Exclusion Criteria:

* Using inhaled corticosteroids
* Pregnant or planning to be pregnant in the next 12 months / Breastfeeding
* Usage of bronchodilators more than three times per week.
* Co-morbidities (as assessed by the primary investigator)
* Taking part in other studies
* Unwilling to withhold bronchodilator, aspirin, anti-coagulant, antihistamine or decongestant medications or caffeine prior to testing procedures.
* FEV1(Forced expiratory volume in one second) < 70% predicted.
* Allergy to lidocaine, fentanyl, midazolam or salbutamol.
* Unstable asthma (i.e exacerbation in 2 weeks preceding testing)

Ages: 19 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Immune response to allergen +/- DE (BAL) | 48 hours
  BAL cellular differential and activation,
Immune response to allergen +/- DE (Th1/Th2/IgE/IgG4) | 48 hours
  Th1/Th2 profile and IgE and IgG4 specific to the allergen used for allergen challenge will be assessed.

SECONDARY OUTCOMES:
Epithelial cell DNA methylation | 48 hours
  Determine if allergen-induced changes in DNA methylation within epithelial cells is augmented by DE (300 µg/m3 inhaled for two hours) and attenuated by PDDE.
Proteomic signature | 48 hours
  Determine if allergen-induced changes in proteomic profile within epithelial cells is augmented by DE (300 µg/m3 inhaled for two hours) and attenuated by PDDE.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Carlsten, MD, MPH, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Calhoun WJ, Jarjour NN, Gleich GJ, Stevens CA, Busse WW. Increased airway inflammation with segmental versus aerosol antigen challenge. Am Rev Respir Dis. 1993 Jun;147(6 Pt 1):1465-71. doi: 10.1164/ajrccm/147.6_Pt_1.1465. PMID 8389107
- [Background] Diaz-Sanchez D, Dotson AR, Takenaka H, Saxon A. Diesel exhaust particles induce local IgE production in vivo and alter the pattern of IgE messenger RNA isoforms. J Clin Invest. 1994 Oct;94(4):1417-25. doi: 10.1172/JCI117478. PMID 7523450
- [Background] Nordenhall C, Pourazar J, Ledin MC, Levin JO, Sandstrom T, Adelroth E. Diesel exhaust enhances airway responsiveness in asthmatic subjects. Eur Respir J. 2001 May;17(5):909-15. doi: 10.1183/09031936.01.17509090. PMID 11488325
- [Result] Carlsten C, Melen E. Air pollution, genetics, and allergy: an update. Curr Opin Allergy Clin Immunol. 2012 Oct;12(5):455-60. doi: 10.1097/ACI.0b013e328357cc55. PMID 22885891
- [Result] Riedl MA, Diaz-Sanchez D, Linn WS, Gong H Jr, Clark KW, Effros RM, Miller JW, Cocker DR, Berhane KT; HEI Health Review Committee. Allergic inflammation in the human lower respiratory tract affected by exposure to diesel exhaust. Res Rep Health Eff Inst. 2012 Feb;(165):5-43; discussion 45-64. PMID 22852485
- [Derived] Robinson A, Huff RD, Ryu MH, Carlsten C. Variants in transient receptor potential channels and toll-like receptors modify airway responses to allergen and air pollution: a randomized controlled response human exposure study. Respir Res. 2023 Sep 7;24(1):218. doi: 10.1186/s12931-023-02518-y. PMID 37679687
- [Derived] Ryu MH, Lau KS, Wooding DJ, Fan S, Sin DD, Carlsten C. Particle depletion of diesel exhaust restores allergen-induced lung-protective surfactant protein D in human lungs. Thorax. 2020 Aug;75(8):640-647. doi: 10.1136/thoraxjnl-2020-214561. Epub 2020 May 28. PMID 32467339
- [Derived] Wooding DJ, Ryu MH, Huls A, Lee AD, Lin DTS, Rider CF, Yuen ACY, Carlsten C. Particle Depletion Does Not Remediate Acute Effects of Traffic-related Air Pollution and Allergen. A Randomized, Double-Blind Crossover Study. Am J Respir Crit Care Med. 2019 Sep 1;200(5):565-574. doi: 10.1164/rccm.201809-1657OC. PMID 30974969